CLINICAL TRIAL: NCT01122797
Title: Study of Metabolism Influence in Human Alcoholic Liver Disease
Brief Title: Influence of Adiponutrin in Chronic Liver Disease
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Eric Trépo, MD, Erasme University Hospital (Olivier Le Moine, MD, PhD)
Other Study IDs: ET-PNPLA3
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2002-12

CONDITIONS: Alcoholic Liver Disease
Keywords: PNPLA3; fibrosis; cirrhosis; alcoholic liver disease
MeSH Terms: conditions — Liver Diseases, Alcoholic; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA extraction from whole blood sample. Piece of liver tissue in the alcoholic liver disease group.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Alcoholic liver disease: Alcoholic liver disease patients undergoing a transjugular liver biopsy in our institution
- Controls: Healthy controls patients recruited from the Occupational Medicine Department during a routine physical examination.

SUMMARY:
Increasing evidence attests the influence of multiple metabolic genetic risk factors in the progression of alcoholic liver disease. Deleterious pathways involved in metabolism such as lipid peroxidation and cytokines have been implicated in promoting inflammation leading to fibrosis increase and liver injury progression. The aim of this study was to assess the role of rs738409 single nucleotide polymorphism in the PNPLA3 gene in alcoholic liver disease patients.

ELIGIBILITY:
ALD patients:

Inclusion Criteria:

* Excess alcohol intake
* Abnormal alanine aminotransferase (ALT) and aspartate aminotransferase (AST) or a suspicion of cirrhosis related to ALD
* Caucasian ethnicity

Exclusion Criteria:

* Presence of any other chronic liver disease
* Co-infection with human immunodeficiency virus

Controls:

Inclusion Criteria:

* Caucasian ethnicity

Exclusion Criteria:

* Presence of a disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing transjugular liver biopsy for alcoholic liver disease will be included in the study to determine the potential correlation between rs738409 PNPLA3 polymorphism and/or PNPLA3 mRNA expression.
Sampling Method: Probability Sample
Enrollment: 658 (Actual)
Dates: Start 2003-01; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Assessment of fibrosis and steatosis by liver biopsy in alcoholic liver disease patients.
  After liver histology assessment for liver liver dammage a potential correlation of fibrosis and steatosis was studied with rs738409 PNPLA3 polymorphism

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Erasme- Dpt of Gastroenterology, Brussels, Belgium

REFERENCES:
- [Background] Tian C, Stokowski RP, Kershenobich D, Ballinger DG, Hinds DA. Variant in PNPLA3 is associated with alcoholic liver disease. Nat Genet. 2010 Jan;42(1):21-3. doi: 10.1038/ng.488. Epub 2009 Nov 29. PMID 19946271
- [Background] Romeo S, Kozlitina J, Xing C, Pertsemlidis A, Cox D, Pennacchio LA, Boerwinkle E, Cohen JC, Hobbs HH. Genetic variation in PNPLA3 confers susceptibility to nonalcoholic fatty liver disease. Nat Genet. 2008 Dec;40(12):1461-5. doi: 10.1038/ng.257. Epub 2008 Sep 25. PMID 18820647
- [Background] Yuan X, Waterworth D, Perry JR, Lim N, Song K, Chambers JC, Zhang W, Vollenweider P, Stirnadel H, Johnson T, Bergmann S, Beckmann ND, Li Y, Ferrucci L, Melzer D, Hernandez D, Singleton A, Scott J, Elliott P, Waeber G, Cardon L, Frayling TM, Kooner JS, Mooser V. Population-based genome-wide association studies reveal six loci influencing plasma levels of liver enzymes. Am J Hum Genet. 2008 Oct;83(4):520-8. doi: 10.1016/j.ajhg.2008.09.012. PMID 18940312
- [Background] Huang Y, He S, Li JZ, Seo YK, Osborne TF, Cohen JC, Hobbs HH. A feed-forward loop amplifies nutritional regulation of PNPLA3. Proc Natl Acad Sci U S A. 2010 Apr 27;107(17):7892-7. doi: 10.1073/pnas.1003585107. Epub 2010 Apr 12. PMID 20385813
- [Background] He S, McPhaul C, Li JZ, Garuti R, Kinch L, Grishin NV, Cohen JC, Hobbs HH. A sequence variation (I148M) in PNPLA3 associated with nonalcoholic fatty liver disease disrupts triglyceride hydrolysis. J Biol Chem. 2010 Feb 26;285(9):6706-15. doi: 10.1074/jbc.M109.064501. Epub 2009 Dec 23. PMID 20034933
- [Background] Kotronen A, Peltonen M, Hakkarainen A, Sevastianova K, Bergholm R, Johansson LM, Lundbom N, Rissanen A, Ridderstrale M, Groop L, Orho-Melander M, Yki-Jarvinen H. Prediction of non-alcoholic fatty liver disease and liver fat using metabolic and genetic factors. Gastroenterology. 2009 Sep;137(3):865-72. doi: 10.1053/j.gastro.2009.06.005. Epub 2009 Jun 12. PMID 19524579
- [Background] Kotronen A, Johansson LE, Johansson LM, Roos C, Westerbacka J, Hamsten A, Bergholm R, Arkkila P, Arola J, Kiviluoto T, Fisher RM, Ehrenborg E, Orho-Melander M, Ridderstrale M, Groop L, Yki-Jarvinen H. A common variant in PNPLA3, which encodes adiponutrin, is associated with liver fat content in humans. Diabetologia. 2009 Jun;52(6):1056-60. doi: 10.1007/s00125-009-1285-z. Epub 2009 Feb 18. PMID 19224197
- [Background] Valenti L, Al-Serri A, Daly AK, Galmozzi E, Rametta R, Dongiovanni P, Nobili V, Mozzi E, Roviaro G, Vanni E, Bugianesi E, Maggioni M, Fracanzani AL, Fargion S, Day CP. Homozygosity for the patatin-like phospholipase-3/adiponutrin I148M polymorphism influences liver fibrosis in patients with nonalcoholic fatty liver disease. Hepatology. 2010 Apr;51(4):1209-17. doi: 10.1002/hep.23622. PMID 20373368
- [Derived] Trepo E, Gustot T, Degre D, Lemmers A, Verset L, Demetter P, Ouziel R, Quertinmont E, Vercruysse V, Amininejad L, Deltenre P, Le Moine O, Deviere J, Franchimont D, Moreno C. Common polymorphism in the PNPLA3/adiponutrin gene confers higher risk of cirrhosis and liver damage in alcoholic liver disease. J Hepatol. 2011 Oct;55(4):906-12. doi: 10.1016/j.jhep.2011.01.028. Epub 2011 Feb 18. PMID 21334404